CLINICAL TRIAL: NCT04982224
Title: A Phase 1/2 Study of REGN5093-M114 (METxMET Antibody-Drug Conjugate) in Patients With MET Overexpressing Advanced Cancer
Brief Title: Study of REGN5093-M114 (METxMET Antibody-Drug Conjugate) in Adult Patients With Mesenchymal Epithelial Transition Factor (MET) Overexpressing Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R5093-M114-ONC-1864; 2020-005065-14 (EudraCT Number)
Record Dates: First submitted 2021-07-20; First posted 2021-07-29 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Advanced NSCLC
Keywords: Non-small cell lung cancer; Mesenchymal epithelial transition factor (MET); MET Overexpressing Advanced Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1. Dose Escalation (Experimental): Cohorts A and B: REGN5093-M114 monotherapy. Cohort C: REGN5093-M114+cemiplimab combination.
  Interventions: Drug: REGN5093-M114; Drug: Cemiplimab
- Phase 2. Dose Expansion (Experimental): Cohorts A and B: REGN5093-M114 monotherapy. Cohort C: REGN5093-M114+cemiplimab combination.
  Interventions: Drug: REGN5093-M114; Drug: Cemiplimab

INTERVENTIONS:
Drug: REGN5093-M114 — Administered by intravenous (IV) infusion
Drug: Cemiplimab — Administered by IV infusion

SUMMARY:
This study is researching an experimental drug called REGN5093-M114 by itself and in combination with cemiplimab. The study is focused on advanced non-small cell lung cancer (NSCLC) that produces too much of a protein called mesenchymal epithelial transition factor (MET) on the cancer cell surface. The aim of the study is to see how safe, tolerable, and effective the study drug is. This study will include 3 study groups, or cohorts, and each group is split into 2 parts:

Part 1: The main purpose of part 1 is to determine a safe dose of REGN5093-M114 (Cohorts A and B), and in combination with cemiplimab (Cohort C).

Part 2: The main purpose of part 2 is to use the REGN5093-M114 dose found for each cohort in part 1 to see how well the study drug works to shrink tumors.

The study is looking at several other research questions, including:

* What side effects may happen from receiving the study drug
* Does the study drug work to reduce or delay the progression of your cancer
* How much study drug is in the blood at different times
* Does the body make antibodies against the study drug (which could make the drug less effective or could lead to side effects)

DETAILED DESCRIPTION:
The trial was intended to be a Phase 1/2 trial, but no participants were enrolled in Phase 2

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed NSCLC that is at advanced stage for which there are no approved therapies available expected to confer clinical benefit as defined in the protocol
2. Willing to provide tumor tissue from newly obtained biopsy from tumor site. Newly obtained biopsies at tissue screening are required. An archival sample can be accepted only after discussion with the medical monitor and if the sample is not more than 6 months old and was obtained on the treatment regimen prior to study screening or after completion of the last therapy. The enrollment of patients will be based on an immunohistochemistry (IHC)-based assay using freshly obtained tumor biopsies or an archival biopsy as described above. Only patients with MET overexpressing tumors by central IHC analysis will be enrolled. For expansion cohorts only: tumor site for biopsy must not have been irradiated previously and must not be the only measurable lesion.
3. Tumor must overexpress MET protein as defined in the protocol
4. For expansion only: At least one lesion that is measurable by RECIST 1.1. Tumor lesions in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions after radiation.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Adequate organ and bone marrow function as defined in the protocol

Key Exclusion Criteria:

1. Has received treatment with an approved systemic therapy or has participated in any study of an investigational agent or investigational device within 2 weeks or 5 half-lives of the prior treatment, whichever is shorter with a minimum of 7 days from the first dose of study therapy
2. Has not yet recovered (ie, grade ≤1 or baseline) from any acute toxicities resulting from prior therapy except as described in the protocol
3. Has received radiation therapy or major surgery within 14 days of first administration of study drug or has not recovered from adverse events as defined in the protocol
4. Another malignancy that is progressing or requires active treatment except as noted in the protocol
5. Untreated or active primary brain tumor, central nervous system (CNS) metastases, leptomeningeal disease, or spinal cord compression as defined in the protocol
6. Encephalitis, meningitis, organic brain disease (eg Parkinson's disease) or uncontrolled seizures in the year prior to first dose of study therapy
7. Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection; or diagnosis of immunodeficiency as defined in the protocol

NOTE: Other protocol-defined Inclusion/ Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) | Up to 28 days
  Dose escalation (Phase 1)
Treatment-emergent adverse events (TEAEs) | Through study completion, an average of 2 years
  Dose escalation (Phase 1)
Serious adverse events (SAEs) | Through study completion, an average of 2 years
  Dose escalation (Phase 1)
TEAEs leading to study treatment discontinuation | Through study completion, an average of 2 years
  Dose escalation (Phase 1)
TEAEs leading to death | Through study completion, an average of 2 years
  Dose escalation (Phase 1)
Laboratory abnormalities (grade 3 or higher per Common Terminology Criteria for Adverse Events [CTCAE]) | Through study completion, an average of 2 years
  Dose escalation (Phase 1)
Concentrations of REGN5093-M114 in serum | Through study completion, an average of 2 years
  Dose escalation (Phase 1)
Total monoclonal antibodies (REGN5093- M114 plus unconjugated antibody) in serum | Through study completion, an average of 2 years
  Dose escalation (Phase 1)
Concentrations of M24 in plasma | Through study completion, an average of 2 years
  Dose escalation (Phase 1)
Concentrations of cemiplimab when given in combination with REGN5093-M114 | Through study completion, an average of 2 years
  Dose escalation (Phase 1) Cohort C
Objective response rate (ORR) | Through study completion, an average of 2 years
  Dose expansion (Phase 2)

SECONDARY OUTCOMES:
ORR | Through study completion, an average of 2 years
  Dose escalation (Phase 1)
TEAEs | Through study completion, an average of 2 years
  Dose expansion (Phase 2)
SAEs | Through study completion, an average of 2 years
  Dose expansion (Phase 2)
TEAEs leading to study treatment discontinuation | Through study completion, an average of 2 years
  Dose expansion (Phase 2)
TEAEs leading to death | Through study completion, an average of 2 years
  Dose expansion (Phase 2)
Laboratory abnormalities (grade 3 or higher per CTCAE) | Through study completion, an average of 2 years
  Dose expansion (Phase 2)
Concentrations of REGN5093-M114 in serum | Through study completion, an average of 2 years
  Dose expansion (Phase 2)
Total monoclonal antibodies (REGN5093- M114 plus unconjugated antibody) in serum | Through study completion, an average of 2 years
  Dose expansion (Phase 2)
Concentrations of M24 in plasma | Through study completion, an average of 2 years
  Dose expansion (Phase 2)
Concentrations of cemiplimab when given in combination with REGN5093-M114 | Through study completion, an average of 2 years
  Dose expansion (Phase 2) Cohort C
Incidence of Anti-drug antibodies (ADA) against cemiplimab over time, when given in combination with REGN5093-M114 | Through study completion, an average of 2 years
  Dose expansion (Phase 2) Cohort C
Titer of ADA against cemiplimab over time, when given in combination with REGN5093-M114 | Through study completion, an average of 2 years
  Dose expansion (Phase 2) Cohort C
Duration of response (DOR) | Through study completion, an average of 2 years
  Phase 1 and Phase 2
Disease control rate (DCR) | Through study completion, an average of 2 years
  Phase 1 and Phase 2
Time to tumor response (TTR) | Through study completion, an average of 2 years
  Phase 1 and Phase 2
Progression free survival (PFS) | Through study completion, an average of 2 years
  Phase 1 and Phase 2
Overall survival (OS) | Through study completion, an average of 2 years
  Phase 1 and Phase 2
Incidence of ADA to REGN5093-M114 over time in monotherapy | Through study completion, an average of 2 years
  Phase 1 and Phase 2
Titer of ADA to REGN5093-M114 over time in monotherapy | Through study completion, an average of 2 years
  Phase 1 and Phase 2
Incidence of ADA to REGN5093-M114 over time in combination with cemiplimab | Through study completion, an average of 2 years
  Phase 1 and Phase 2
Titer of ADA to REGN5093-M114 over time in combination with cemiplimab | Through study completion, an average of 2 years
  Phase 1 and Phase 2

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (11):
- United States (11):
  - University of California Irvine School of Medicine - Suite 400, Room 407, Orange, California
  - University of Colorado Hospital Anshutz Outpatient Pavillion, Denver, Colorado
  - Johns Hopkins Hospital - Clinical Study Location - Skip Viragh Outpatient Cancer Building, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center - 4F Second Medical Building, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Henry Ford Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pittsburgh Medical Center - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Next Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/